CLINICAL TRIAL: NCT06801951
Title: Effects of Oral Nutritional Supplement and Acute Resistance Exercise in Chronic Obstructive Pulmonary Disease
Brief Title: Oral Supplement and Acute Resistance Exercise
Acronym: HMB exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0655
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: oral nutrition supplement; resistance exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EAA + HMB (Experimental): Targeted amino acid formulation (7.0 g EAA and 1.5 g HMB (EAA+HMB))
  Interventions: Other: acute resistance exercise with oral nutrition supplementation; Other: stable tracer infusion
- Placebo (Placebo Comparator): 7.0 gram non-essential amino acids
  Interventions: Other: acute resistance exercise with oral nutrition supplementation; Other: stable tracer infusion

INTERVENTIONS:
Other: acute resistance exercise with oral nutrition supplementation — acute bout of resistance exercise on an isokinetic exercise machine of each limb (i.e., right and left arm and right and left leg) allowing control of velocity and force. Immediately upon completion, 1 serving of liquid nutrition supplement will be consumed. An additional serving of the liquid nutrition supplement will be sent home for consumption in the evening.
Other: stable tracer infusion — stable isotopes Such as L-[ring-13C6]-Phenylalanine, L-[ring-D4]Tyrosine, L-[Methyl-D3]Tau-Methylhistidine, trans-[2,5,5-D3]4-Hydroxy-L-proline, L-[Guanido-15N2]-Arginine, L-[4,4,5,5-D4-5-13C]Citruline, L-13C5 -Ornithine, L-15N2-Glutamine, L-[1,2-13C2]Glutamic Acid, 1-13C-Glycine, L-15N3-Histidine, L-13C6-Leucine, L-[methyl-D3]Methionine, α-1-13C-ketoisocaproic acid, L-1-13C-Methionine, DL-[3,3,4,4-D4]Homocysteine, L-[1,2-13C2]Taurine, L-(Indole-D5)Tryptophan, 13C-Urea, L-1-13C-Isoleucine, L-13C5-Valine, α-[Dimethyl-13C2]ketoisovaleric acid, 2-keto-3-methyl-13C6-pentanoate, 3-hydroxy-[3,4-methyl-13C3]isovaleric acid, 13C3-glycerol is given IV simultaneously

SUMMARY:
This study should provide the mechanistic basis for and evaluation of a new nutritional formulation to be used alongside exercise training to improve muscle function and exercise performance by minimizing exercise induced metabolic deregulation in patients with Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
Our central hypothesis is that improving the metabolic response to resistance exercise via targeted nutritional modulation with EAA enriched with HMB (EAA+HMB) will increase the gain in muscle function and exercise performance by positively influencing skeletal muscle protein homeostasis among severe COPD patients. Our rationale for the proposed research is that detailed insight in the mechanisms by which resistance exercise induces metabolic deregulations in severe COPD patients, and demonstration of the effectiveness of targeted nutritional intervention will provide opportunities for the development of innovative safe and effective nutritional approaches to improve their training response and skeletal muscle repair, leading to increased daily life physical activity. Furthermore, the proposed studies will provide supportive data of, and focus for a subsequent phase 2b/3 clinical trial to improve quality of life, and clinical outcomes of severe COPD patients. We propose to study simultaneously the following specific aim:

Investigate the metabolic mechanisms by which resistance exercise induces protein catabolism in severe COPD patients as compared to healthy age and gender matched control subjects. Our working hypothesis is that patients with severe COPD (GOLD II-IV) have a metabolic signature that relates to their late (24h) post-exercise catabolic response. We will utilize an innovative IV tracer pulse approach of > 15 labeled amino acids to enable kinetic analysis of their intracellular production, disposal and interconversion rates (fluxomics), and quantify the rates of muscle protein synthesis and breakdown.

The liquid nutrition supplement will be either targeted amino acid formulation (7.0 g EAA and 1.5 g HMB (EAA+HMB)) or placebo (7.0 gram non-essential amino acids). Liquid nutrition supplement will be given to subjects according to a randomized, placebo controlled, double blind, cross-over design.

ELIGIBILITY:
Inclusion criteria COPD subjects:

Ability to walk, sit down and stand up independently

Age 45 - 100 years

Willing to lay in bed for 4 hours during study visits

Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: FEV1 < 70% of reference FEV1

Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day

Shortness of breath on exertion

Willingness and ability to comply with the protocol

Inclusion criteria control subjects:

Healthy male or female according to the investigator's or appointed staff's judgment

Ability to walk, sit down and stand up independently

Age 45 - 100 years

Willing to lay in bed for 4 hours during long study visits

No diagnosis of COPD

Willingness and ability to comply with the protocol

Exclusion Criteria all subjects:

Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (healthy subjects only)

Subjects 86 years and older that fail to get physician eligibility confirmation

Established diagnosis of Insulin dependent diabetes mellitus

Established diagnosis of malignancy

History of untreated metabolic diseases including hepatic or renal disorder

Presence of acute illness or metabolically unstable chronic illness

Presence of fever within the last 3 days

Use of short course of oral corticosteroids within 4 weeks preceding study day

Dietary or lifestyle characteristics:

Use of protein or amino acid containing nutritional supplements within 5 days of first test day

Indications related to interaction with study products:

Known allergy or sensitivity to milk or milk products

Previous injury that could interfere with participation in resistance exercise protocol

Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

(Possible) pregnancy

Already enrolled in another clinical trial and that clinical trial interferes with participating in this study

Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient

Ages: 45 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
net whole body protein metabolism synthesis | 2, 5, 10, 15, 20, 30, 40, 50, 60, 90, 120, 150, 180, 210 and 240 ± 5 minutes
  Change in whole-body protein synthesis rate and myofibrillar protein breakdown

CONTACTS AND LOCATIONS:
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No